CLINICAL TRIAL: NCT03183947
Title: Symptom Based Treatment Affects Brain Plasticity - Cognitive Training in Patients With Affective Symptoms
Acronym: APIC-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-094
Record Dates: First submitted 2017-06-02; First posted 2017-06-12 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Depression; Schizophrenia
Keywords: fMRI; neurofeedback; emotion regulation; schizophrenia; cognitive reappraisal; depression
MeSH Terms: conditions — Depression; Schizophrenia; Emotional Regulation | interventions — Neurofeedback; Gene Expression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fMRI Neurofeedback regulation of left PFC (Experimental): Study related procedures included: PANAS, BDI-II, ERQ (questionnaires or evaluations)
  Interventions: Procedure: fMRI; Behavioral: Neurofeedback; Other: PANAS; Other: BDI-II; Other: ERQ
- fMRI Neurofeedback of right PFC (Experimental): Study related procedures included: PANAS, BDI-II, ERQ (questionnaires or evaluations)
  Interventions: Procedure: fMRI; Behavioral: Neurofeedback; Other: PANAS; Other: BDI-II; Other: ERQ

INTERVENTIONS:
Procedure: fMRI — collection of functional brain data for 1 hour per day
  Other Names: functional magnetic resonance imaging
Behavioral: Neurofeedback — Task of the participants is to increase the activity in the selected brain region (left or right prefrontal cortex). After regulation they will get a feedback about the regulation success. (Patients: days 3 & 4; controls: Days 2 & 3)
Other: PANAS — to assess the mood before and after the fMRI and after 4 weeks during a telephone interview
  Other Names: Positive And Negative Affect Scales
Other: BDI-II — to assess depressive symptomatology before neurofeedback and 4 weeks after the intervention during telephone interview
  Other Names: Beck's depression inventory
Other: ERQ — To assess emotion regulation strategies before and after neurofeedback training (patients: day 3&4; controls: day 2&3) and after 4 weeks during a telephone interview
  Other Names: Emotion regulation questionnaire

SUMMARY:
The aim of the study is the examination of brain plasticity on on affective symptoms after neuromodulation with fMRI (functional magnetic resonance imaging) neurofeedback. During the fMRI neurofeedback training, patients with depression as well as patients with schizophrenia are trained to consciously regulate the activity of areas which are associated with the cognitive reappraisal of emotional stimuli.The aim is to improve the patients' subjective emotional processing and perception in everyday life as well as to investigate the impact of neurofeedback on resting-state networks in the brain. Healthy participants will be investigated as control group.

DETAILED DESCRIPTION:
The ability to regulate emotions is a central element of mental health that is significantly affected in various psychiatric disorders. Its importance for development and maintenance of depressive symptomatology has been widely shown; e.g. patients with depression have a significantly reduced ability to regulate emotions in response to negative stimuli. However, emotion regulation abilities may pose as an important resilience factor that can counteract the development of depressive symptoms. The loss of the ability to regulate emotions is not only observed in depression, but is also a core factor in negative symptoms of schizophrenia.

Cognitive reappraisal training is an established method to improve emotion regulation. The cognitive reappraisal of a stimulus or situation works by reinterpreting the emotional stimulus or situation and can change the course of the emotional response. Over the last years this form of cognitive reappraisal training has become a standard approach in the treatment of affective disorders.

The prefrontal cortex (PFC) plays an important role in emotion regulation. In line with this it has been shown that patients with reduced emotion regulation ability display impaired functioning of the PFC. Aim of the study is to train patients to consciously upregulate activity in the PFC and thereby to increase emotion regulation ability. On the behavioral level this is expected to correlate with a reduced experience of negative mood. In order to regulate the PFC, participants are instructed to use cognitive reappraisal strategies. Cognitive reappraisal is an effective and well-investigated strategy to improve emotion regulation and is a standard cognitive-behavioral psychotherapeutic intervention. During cognitive reappraisal the meaning of a picture is reinterpreted in order to reduce the emotional reaction. Recent fMRI studies have shown that cognitive reappraisal is associated with an increase in prefrontal activity and a decrease of amygdala activation.

The new technique of real-time fMRI enables subjects to influence their brain activity in certain areas based on neurofeedback. Ongoing brain activity as measured by fMRI is reported to the participants in real time via brain computer interface (BCI). In order to influence brain activity, mental strategies are usually recommended to the participants that have been shown to increase activity in the respective area. Due to the identification of contingency between feedback and mental strategies participants are able to control their own brain activity consciously. It has been shown that psychiatric symptomatology can be improved using this non-invasive technique. In the current study it will be investigated whether neurofeedback of the PFC has a positive influence on affective symptoms in patients with depression and schizophrenia, respectively. In detail it is researched whether the upregulation of activity in the PFC can lead to an increase in subjective well-being. Two groups of patients (depression (N=40) and schizophrenia (N=40)) as well as a group of healthy participants will receive neurofeedback-training of the PFC. Aim of the study is an improvement of depressive (or negative) symptoms as well as the investigation of the impact of neurofeedback on resting-state networks in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Depression according to ICD-10 (F32.x, F33.x, F31.3 or F34.x); Schizophrenia according to ICD-10 (F2x); or healthy subjects
* Fluent German language skills

Exclusion Criteria:

* any contraindication to MRI examination or claustrophobia
* pregnant or lactating women
* acute suicidal tendency
* persons incapable of giving consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
change in self-control over neuronal activity in PFC | 1 week
  fMRI-BCI as a measure before and after the regulation of the brain activity

SECONDARY OUTCOMES:
Changes from baseline in brain plasticity | 2 weeks
  fMRI as a measure for brain plasticity before and after neurofeedback
Change in pathology (depression) | 4 weeks after interventions
  BDI-II as a measure of the intensity and quality of depressive symptoms before training and 4 weeks following the intervention
specificity of left or right PFC neurofeedback | 2 weeks
change in resting state brain activation | 2 weeks
  Resting state fMRI as a measure before and after neurofeedback
Change in pathology (mood) | 4 weeks after interventions
  Positive And Negative Affect Scales (PANAS) as a measure of mood before and after the fMRI and after 4 weeks during a telephone interview

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Mathiak, Prof MD PhD, Principal Investigator — University Hospital RWTH Aachen, Department of Psychiatry, Psychotherapy and Psychosomatics
Locations (1):
- University Hospital RWTH Aachen, Department of Psychiatry, Psychotherapy and Psychosomatics, Aachen, Germany

REFERENCES:
- [Background] Buhle JT, Silvers JA, Wager TD, Lopez R, Onyemekwu C, Kober H, Weber J, Ochsner KN. Cognitive reappraisal of emotion: a meta-analysis of human neuroimaging studies. Cereb Cortex. 2014 Nov;24(11):2981-90. doi: 10.1093/cercor/bht154. Epub 2013 Jun 13. PMID 23765157
- [Background] Hayes JP, Vanelzakker MB, Shin LM. Emotion and cognition interactions in PTSD: a review of neurocognitive and neuroimaging studies. Front Integr Neurosci. 2012 Oct 9;6:89. doi: 10.3389/fnint.2012.00089. eCollection 2012. PMID 23087624
- [Background] Kohn N, Eickhoff SB, Scheller M, Laird AR, Fox PT, Habel U. Neural network of cognitive emotion regulation--an ALE meta-analysis and MACM analysis. Neuroimage. 2014 Feb 15;87:345-55. doi: 10.1016/j.neuroimage.2013.11.001. Epub 2013 Nov 9. PMID 24220041
- [Background] Linden DE, Habes I, Johnston SJ, Linden S, Tatineni R, Subramanian L, Sorger B, Healy D, Goebel R. Real-time self-regulation of emotion networks in patients with depression. PLoS One. 2012;7(6):e38115. doi: 10.1371/journal.pone.0038115. Epub 2012 Jun 4. PMID 22675513
- [Background] Ochsner KN, Bunge SA, Gross JJ, Gabrieli JD. Rethinking feelings: an FMRI study of the cognitive regulation of emotion. J Cogn Neurosci. 2002 Nov 15;14(8):1215-29. doi: 10.1162/089892902760807212. PMID 12495527
- [Background] Weiskopf N, Scharnowski F, Veit R, Goebel R, Birbaumer N, Mathiak K. Self-regulation of local brain activity using real-time functional magnetic resonance imaging (fMRI). J Physiol Paris. 2004 Jul-Nov;98(4-6):357-73. doi: 10.1016/j.jphysparis.2005.09.019. Epub 2005 Nov 10. PMID 16289548
- [Background] Joormann J, Gotlib IH. Emotion regulation in depression: relation to cognitive inhibition. Cogn Emot. 2010 Feb 1;24(2):281-98. doi: 10.1080/02699930903407948. PMID 20300538
- [Background] Troy AS, Wilhelm FH, Shallcross AJ, Mauss IB. Seeing the silver lining: cognitive reappraisal ability moderates the relationship between stress and depressive symptoms. Emotion. 2010 Dec;10(6):783-95. doi: 10.1037/a0020262. PMID 21058843
- [Derived] Keller M, Zweerings J, Klasen M, Zvyagintsev M, Iglesias J, Mendoza Quinones R, Mathiak K. fMRI Neurofeedback-Enhanced Cognitive Reappraisal Training in Depression: A Double-Blind Comparison of Left and Right vlPFC Regulation. Front Psychiatry. 2021 Aug 23;12:715898. doi: 10.3389/fpsyt.2021.715898. eCollection 2021. PMID 34497546